CLINICAL TRIAL: NCT03006263
Title: Randomized Controlled Trials on Clinical Outcomes of Totally Laparoscopic Versus Laparoscopy Assisted Total Gastrectomy for Gastric Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Professor, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2016YF021-02
Record Dates: First submitted 2016-12-26; First posted 2016-12-30 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms; Totally Laparoscopic Total Gastrectomy; Laparoscopy Assisted Total Gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Totally Laparoscopic Total Gastrectomy (Experimental): Totally Laparoscopic Total Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Totally Laparoscopic Total Gastrectomy
- Laparoscopy Assisted Total Gastrectomy (Experimental): Laparoscopy Assisted Total Gastrectomy will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: Laparoscopy Assisted Total Gastrectomy

INTERVENTIONS:
Procedure: Totally Laparoscopic Total Gastrectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy,Totally Laparoscopic Total Gastrectomy will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience.
  Arms: Totally Laparoscopic Total Gastrectomy
Procedure: Laparoscopy Assisted Total Gastrectomy — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy,Laparoscopy Assisted Total Gastrectomy will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience.
  Arms: Laparoscopy Assisted Total Gastrectomy

SUMMARY:
The purpose of this study is to explore clinical outcomes of totally laparoscopic versus laparoscopy assisted total gastrectomy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 75 years old
2. Primary gastric adenocarcinoma (papillary, tubular, mucinous, signet ring cell, or poorly differentiated) confirmed pathologically by endoscopic biopsy
3. Locally advanced tumor in the middle third stomach（cT1-4a, N-/+, M0 at preoperative evaluation according to the AJCC(American Joint Committee on Cancer) Cancer Staging Manual Seventh Edition）
4. No distant metastasis, no direct invasion of pancreas, spleen or other organs nearby in the preoperative examinations
5. Performance status of 0 or 1 on ECOG (Eastern Cooperative Oncology Group) scale
6. ASA (American Society of Anesthesiology) class I to III
7. Written informed consent

Exclusion Criteria:

1. Pregnant and lactating women
2. Suffering from severe mental disorder
3. History of previous upper abdominal surgery (except for laparoscopic cholecystectomy)
4. History of previous gastric surgery (including ESD/EMR (Endoscopic Submucosal Dissection/Endoscopic Mucosal Resection )for gastric cancer)
5. Enlarged or bulky regional lymph node （diameter over 3cm）supported by preoperative imaging including enlarged or bulky No.10 lymph node
6. History of other malignant disease within the past 5 years
7. History of previous neoadjuvant chemotherapy or radiotherapy
8. History of unstable angina or myocardial infarction within the past 6 months
9. History of cerebrovascular accident within the past 6 months
10. History of continuous systematic administration of corticosteroids within 1 month
11. Requirement of simultaneous surgery for other disease
12. Emergency surgery due to complication (bleeding, obstruction or perforation) caused by gastric cancer
13. FEV1<50% of the predicted values

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2021-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
overall postoperative morbidity rates | 30 days
  Refers to the incidence of early postoperative complications. The early postoperative complication are defined as the event observed within 30 days after surgery.

SECONDARY OUTCOMES:
3-year overall survival rate | 36 months
3-year disease free survival rate | 36 months
3-year recurrence pattern | 36 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.
Intraoperative morbidity rates | 1 day
  The intraoperative postoperative morbidity rates are defined as the rates of event observed within operation.
Time to first ambulation | 30 days
  Time to first ambulation in hours is used to assess the postoperative recovery course.
Time to first flatus | 30 days
  Time to first flatus in days is used to assess the postoperative recovery course.
Time to first liquid diet | 30 days
  Time to first liquid diet in days is used to assess the postoperative recovery course.
Time to first soft diet | 30 days
  Time to first soft diet in days is used to assess the postoperative recovery course.
Duration of postoperative hospital stay | 30 days
  Duration of postoperative hospital stay in days is used to assess the postoperative recovery course.
Postoperative pain | 30 days
  Visual analog pain score method is used to evaluate the difference of postoperative pain degree.The score of postoperative pain is used to assess the postoperative recovery course.
The variation of weight | 3, 6, 9 and 12 months
  The variation of weight on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The variation of cholesterol | 3, 6, 9 and 12 months
  The variation of cholesterol in millimole/liter on postoperative 3, 6, 9 and 12 months are used to access the postoperative nutritional status and quality of life.
The results of endoscopy | 3 and 12 months
  The incidence of reflux esophagitis under the endoscopy on postoperative 3 and 12 months are used to access the postoperative quality of life.
The variation of body temperature | 8 days
  The daily highest body temperature in degree centigrade before discharge are recorded to access the inflammatory and immune response.
The variation of white blood cell count | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of white blood cell count from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of hemoglobin | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of hemoglobin in gram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.
The variation of C-reactive protein | Preoperative 3 days and postoperative 1, 3, and 5 days
  The values of C-reactive protein IN milligram/liter from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded to access the inflammatory and immune response.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, Professor, Principal Investigator — Fujian Medical University Union Hospital,China

IPD SHARING:
Plan to Share IPD: No